CLINICAL TRIAL: NCT05574374
Title: A Randomized, Open-label, Three-sequence, Three-period, Multiple Dosing Crossover, Phase 1 Clinical Trial to Evaluate the Effect of DWP14012 on the Pharmacodynamics of DWC202202 in Combination With DWP14012 in Healthy Subjects
Brief Title: Drug-drug Interactions Between DWP14012 and DWC202202 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP14012110
Record Dates: First submitted 2022-09-04; First posted 2022-10-10 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — fexuprazan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): * Treatment A: DWC202202 1 tablet qd for 7days
  * Treatment B: DWC202202 1 tablet qd + DWP14012 1 tablet qd for 7days
  * Treatment C: DWC202202 1 tablet qd + DWC202203 1 tablet qd for 7days
  Interventions: Drug: DWP14012; Drug: DWC202202; Drug: DWC202203
- Cohort 2 (Experimental): * Treatment C: DWC202202 1 tablet qd + DWC202203 1 tablet qd for 7days
  * Treatment A: DWC202202 1 tablet qd for 7days
  * Treatment B: DWC202202 1 tablet qd + DWP14012 1 tablet qd for 7days
  Interventions: Drug: DWP14012; Drug: DWC202202; Drug: DWC202203
- Cohort 3 (Experimental): * Treatment B: DWC202202 1 tablet qd + DWP14012 1 tablet qd for 7days
  * Treatment C: DWC202202 1 tablet qd + DWC202203 1 tablet qd for 7days
  * Treatment A: DWC202202 1 tablet qd for 7days
  Interventions: Drug: DWP14012; Drug: DWC202202; Drug: DWC202203

INTERVENTIONS:
Drug: DWP14012 — Potassium-competitive acid blocker
Drug: DWC202202 — Clopidogrel Bisulfate
Drug: DWC202203 — Proton pump inhibitor

SUMMARY:
A randomized, open-label, three-sequence, three-period, multiple dosing crossover, phase 1 clinical trial to evaluate the effect of DWP14012 on the pharmacodynamics of DWC202202 in combination with DWP14012 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥ 19 and ≤ 50 years at screening
* Subjects with a body weight ≥ 50.0 kg to ≤ 90.0 kg with a body mass index (BMI) of ≥ 18.0 kg/m2 to ≤ 27.0 kg/m2 at screening

  ※ BMI (kg/m2) = body weight (kg)/[height (m)]2
* Subjects who voluntarily decided to participate in the study and provided written consent to follow precautions after receiving a sufficient explanation on this study and fully understanding the information
* Subjects who are eligible to participate in the study at the discretion of the investigator by physical examination, laboratory tests, and investigator questioning, etc.

Exclusion Criteria:

* Subjects with a history related to blood clotting disorder or bleeding
* Subjects with hypersensitivity or history of clinically significant hypersensitivity to drugs including potassium competitive acid blocker [P-CAB] class, aspirin, antibiotics, etc.
* Subjects with a history of drug abuse or a positive result of using abusive drugs in the urine drug screen
* Subjects who participated in other clinical trials (including bioequivalence studies) within 6 months prior to the first scheduled dose of the IP
* Subjects who donated whole blood within 2 months, donated blood components within 1 month, or received blood transfusion within 1 month prior to the first scheduled dose
* Subjects who are unable to refrain from grapefruit-containing products from 3 days prior to the first scheduled dose until last discharge from hospital
* Subjects with hereditary disorders including galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, etc.
* Subjects or their spouses or partners who are unable to use medically acceptable appropriate double-method of contraception or medically acceptable contraception throughout the study period and for at least 4 weeks after the last IP administration
* Subjects who are smoking

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Emax | up to 50 days
AUEC0-24 | up to 50 days

SECONDARY OUTCOMES:
DWC202202 Cmax,ss | up to 50 days
DWC202202 active metabolite Cmax,ss | up to 50 days
DWC202202 AUCtau,ss | up to 50 days
DWC202202 active metabolite AUCtau,ss | up to 50 days
DWC202202 AUCinf,ss | up to 50 days
DWC202202 active metabolite AUCinf,ss | up to 50 days
DWC202202 Tmax,ss | up to 50 days
DWC202202 active metabolite Tmax,ss | up to 50 days
DWC202202 t1/2,ss | up to 50 days
DWC202202 active metabolite t1/2,ss | up to 50 days
DWC202202 Cmin,ss | up to 50 days
DWC202202 active metabolite Cmin,ss | up to 50 days
DWC202202 Cavg,ss | up to 50 days
DWC202202 active metabolite Cavg,ss | up to 50 days
DWC202202 CLss/F | up to 50 days
DWC202202 Vd,ss/F | up to 50 days
DWC202202 PTF (peak to trough fluctuation) | up to 50 days
DWC202202 active metabolite PTF (peak to trough fluctuation) | up to 50 days
DWC202202 R | up to 50 days
DWC202202 active metabolite MR | up to 50 days

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided